CLINICAL TRIAL: NCT01015300
Title: D0904 - A Pilot Study of Bevacizumab (Avastin) in Patients With Unresectable or Recurrent Hemangioblastoma From Von Hippel-Lindau Disease.
Brief Title: Bevacizumab (Avastin) in Unresectable/Recurrent Hemangioblastoma From Von-Hippel-Lindau Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study terminated due to low accrual.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0904
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Hemangioblastomas; Von Hippel Lindau Disease
Keywords: Hemangioblastoma; Von Hippel Lindau; VHL; lesion; EGFR
MeSH Terms: conditions — Hemangioblastoma; von Hippel-Lindau Disease | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Avastin — Patients will receive Bevacizumab (Avastin) 10mg/kg IV every two weeks for 6 months

SUMMARY:
Von Hippel-Lindau (VHL) disease is an inherited syndrome manifested by a variety of benign and malignant tumors. Hemangioblastomas are the most common lesion associated with VHL disease affecting 60-84% of patients with a mean age at diagnosis of 29 years. Standard treatment for this disease is by surgery or radiotherapy. No approved systemic therapy yet exists. Patients with VHL have an increased growth factor production, specifically vascular endothelial growth factor (VEGF), resulting in angiogenesis (growth of blood vessels). Studies show that Bevacizumab inhibits the growth of VEGF protein and will block the VEGF-driven angiogenesis and result in stabilization and regression of hemangioblastomas in VHL disease patients. The dose of bevacizumab will be 10 mg/kg every two weeks for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* One or more CNS hemangioblastomas not amendable to surgical resection or recurrent post resection
* Confirmed diagnosis of von-Hippel-Lindau disease
* No prior treatment with VEGF inhibitors
* Index hemangioblastomas lesion at least 5mm on MRI
* No major bleeding event from hemangioblastoma within 90 days
* KPS > or equal to 60%
* Age > or equal to 18 years

Exclusion Criteria:

* Prior treatment with VEGF inhibitors
* Major bleeding event from hemangioblastoma within 90 days
* Inability to comply with study and/or follow up procedures
* Life expectancy of less than 12 weeks
* Current or recent (within 4 weeks of the first infusion of this study) participation in an experimental drug study other than a Genentech sponsored bevacizumab cancer study
* Active malignancy will be permissible if treating physician deems that concurrent administration of bevacizumab is not contraindicated and that the patient would be able to complete with the other parameters of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Radiographic response in the size of the hemangioblastoma on magnetic resonance imaging (MRI) | 24 months

SECONDARY OUTCOMES:
Changes in VEGF with bevacizumab treatment assist in the predication of radiographic response. Products of the HIF-1A synthesis pathway: plasma VEGF, PDGF, TGF-a and erythropoietin. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: J Marc Pipas, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States